CLINICAL TRIAL: NCT03947502
Title: Effectiveness of a Structured Group Intervention Based on Pain Neuroscience Education for Patients With Fibromyalgia in Primary Care: a Multicenter Randomized Open-label Controlled Trial
Brief Title: Pain Neuroscience Education as Treatment in Fibromyalgia Affected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osatzen Sociedad Vasca Medicina Familiar y Comunitaria (Other)
Responsible Party: Principal Investigator, maría muñoa capron-manieux, Head of Primary Care Setting (Alango), Osatzen Sociedad Vasca Medicina Familiar y Comunitaria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2016097 (SO)
Record Dates: First submitted 2019-05-01; First posted 2019-05-13 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; pain; neurobiology; education; movement
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Intervention Model Description: Multicentre (5 nodes) randomized clinical trial, Pain neuro education based on 6 weekly classes of 2 hours for patients affected by fibromyalgia, taught by a multidisciplinary group. Controlled with usual therapies treated group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group with (Experimental): Educational intervention in neurobiology of pain
  Interventions: Behavioral: Educational intervention in neurobiology of pain
- Control group (No Intervention): The control group is treated with usual medication for fibromyalgia, anxiolytics, antidepressants, analgesics, ... Depending on the medical needs and criteria of patients´s primary care physician.

INTERVENTIONS:
Behavioral: Educational intervention in neurobiology of pain — The educational intervention will intend to make the individual aware that in the processes of learning, sensitization, habituation and acquisition of beliefs about pain there are automatic unconscious mechanisms, which can be modulated through conscious behaviors. Based on this the investigators propose the active participation of patients in the process of desensitization of their central nervous system. The investigators will try to encourage attention and weaken the neuronal connections that make up the pain neuromatrix to establish new connections thanks to neuroplasticity.
  Arms: Intervention Group with

SUMMARY:
Fibromyalgia (FM) is a chronic, complex and disabling clinical entity that has an average global prevalence of 2.7%. It occurs mainly in women in a 3: 1 ratio. It is characterized by persistent generalized pain, fatigue, unrefreshing sleep, cognitive dysfunction and numerous systemic symptoms such as dizziness, migraine, digestive alterations or sensory intolerances. At present there is no pharmacological treatment with specific indication for fibromyalgia. Usually, non-curative treatments are recommended that alleviate the symptoms of the patients and improve their quality of life and functionality.

The investigator's main goal is to evaluate the effectiveness at 1 year of a group educational intervention in neurobiology of pain in patients affected by fibromyalgia, in comparison with the evolution of a control group that will continue only with its usual treatments. This intervention will be carried out in the field of Primary Care and its effectiveness will be assessed by reducing or not having diagnostic criteria (reduction of areas of pain and of the severity of fibromyalgia symptoms), using the Criteria for the Diagnosis of Fibromyalgia of the American College of Rheumatology 2010 (ACR 2010).

DETAILED DESCRIPTION:
Methodology of the project In group sessions of 14 patients, a health professional explained the neurological mechanisms that are behind the perception of pain, fatigue and illness from the recent knowledge in neuroscience about brain and pain, as well as the brain's ability to change patien´s behaviour thanks to neuroplasticity.

There will be 5 sessions of 2 hours per week and another one per month. Before the latter, a workshop of 2 hours of movement will be given.

Each week the contents of the class and other complementary materials will be sent to the patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of fibromyalgia stablished by the American Rheumatology College criteria 2010,
* Older than 18 years
* Have signed the informed consent

Exclusion Criteria:

* Psychiatric or neurological disorder which could prevent assimilate the training
* Refusal to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
To asses the number of patients that stop fulfilling fibromyalgia criteria (American College of Reumathology 2010 criteria). | It will be measured at 12-months after the beginning of the intervention,
  The criteria established by the American College of Reumathology 2010 will be measured to estimate the negativization of the fibromyalgia diagnostic criteria. (Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Ménard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovský J, Wolfe F, Hawker G. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010 Sep;62(9):2569-81. doi: 10.1002/art.27584. PubMed PMID: 20872595.

SECONDARY OUTCOMES:
To asses the effectiveness by modified- PNE to improve fibromyalgia symptoms and security; meassured by effecte size and group intervention time size. | It will be measured at 1 month, 6 months and 12-months after the beginning of the intervention,
  Fibromyalgia Impact Questionnaire: is composed of 10 questions. It measures the functionality of patients with fibromyalgia. 0-100 and 100 the worst.
To asses the decrease in pain by modified- PNE to improve fibromyalgia symptoms and security; meassured by effecte size and group intervention time size. | t will be measured at 1 month, 6 months and 12-months after the beginning of the intervention,
  Brief Pain Inventory: it measures pain. The most point the worst (0-100).
To assesthe decrease in catastrophising by modified- PNE to improve fibromyalgia symptoms and security; meassured by effecte size and group intervention time size. | t will be measured at 1 month, 6 months and 12-months after the beginning of the intervention,
  Pain catastrophising scale: it measures catastrophizing. The most point the worst (0-100).
To asses the decrease in anxiety and depression by modified- PNE to improve fibromyalgia symptoms and security; meassured by effecte size and group intervention time size. | t will be measured at 1 month, 6 months and 12-months after the beginning of the intervention,
  Hospital Anxiety and Depression scale: 0-7 = Normal; 8-10 = Borderline 11-21 = Abnormal.
To asses the security of modified- PNE to improve fibromyalgia symptoms and security; meassured by effecte size and group intervention time size. | It will be measured at 12-months after the beginning of the intervention,
  Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v4.0.